CLINICAL TRIAL: NCT00565721
Title: A Phase 2, Open-label, Proof-of-concept Study to Assess the Ability to Detect Tumours and Angiogenesis Via the Expression of ανβ3/5 Integrin Receptors by [18F]AH-111585 PET Imaging
Brief Title: A Proof-of-concept Study to Assess the Ability of [18F]AH-111585 PET Imaging to Detect Tumours and Angiogenesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-135-003; NCT00923767 (obsolete NCT alias)
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: High-grade Glioma; Lung Cancer; Head & Neck Cancer; Sarcoma; Melanoma
Keywords: Static PET imaging; Dynamic PET imaging; Angiogenesis; αvβ3 integrins; oncology imaging
MeSH Terms: conditions — Glioma; Lung Neoplasms; Head and Neck Neoplasms; Sarcoma; Melanoma | interventions — AH 111585

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluciclatide Injection - (AH111585 (F18)) (Experimental): Using of the drug product named, AH111585 (F18) Injection. It's generic chemical name is Fluciclatide.
  Interventions: Drug: Fluciclatide Injection - (AH111585 (F18))

INTERVENTIONS:
Drug: Fluciclatide Injection - (AH111585 (F18)) — 18F labelled Cyclic RGD peptide PET agent for injection.
  Other Names: Fluciclatide

SUMMARY:
This proof-of-concept study is designed to assess the ability of [18F]AH-111585 PET imaging to detect tumors and angiogenesis. Up to 30 evaluable subjects are planned to be included at up to 2 study centers in the US. Subjects are considered evaluable if they undergo administration of AH-111585 (18F) Injection, dynamic and static PET imaging, and tumor tissue acquisition. The targeted population is adult subjects at initial diagnosis or recurrence with tumors ≥2.5 cm in diameter who are scheduled to undergo resection or biopsy of the tumor as a result of routine clinical treatment. The tumors must belong to one of the following 5 types:

* High-grade glioma, including glioblastoma multiforme, anaplastic astrocytoma, and anaplastic oligodendroglioma
* Lung cancer, including small cell lung cancer and non-small cell lung cancer
* Head and neck (H&N) tumors, including laryngeal squamous cell carcinoma, well-differentiated thyroid and oral cavity carcinoma
* Sarcoma
* Melanoma

Safety will be assessed from the rates of adverse events, changes in vital signs, changes in electrocardiogram (ECG) parameters, changes in physical examination findings, and changes in clinical laboratory findings.

Efficacy will be assessed as the correlations between parameters derived from the PET images and the reference standards. The reference standards will be immunohistology for αvβ3 integrins and other biomarkers specific for oncology and angiogenesis and from the standard of care imaging.

Measures obtained from optional DCE-CT imaging may also be used to compare the uptake and retention of [18F]AH-111585 in tumors obtained from the dynamic PET to assess functional status of the vascular system of the tumor.

ELIGIBILITY:
Selection of Subjects: The targeted subject population is adult subjects at initial diagnosis or recurrence with tumours ≥2.5 cm in diameter who are scheduled to undergo resection or biopsy of the tumour as a result of routine clinical treatment.

General Inclusion Criteria for all Subjects:

* The subject is ≥18 years old.
* The subject has been diagnostically imaged and is suspected of having a primary or metastatic tumour lesion ≥2.5 cm of one of the following types: high-grade glioma, including glioblastoma multiforme, anaplastic astrocytoma, and anaplastic oligodendroglioma; lung cancer, including small cell lung cancer and non-small cell lung cancer; H&N tumours, including laryngeal squamous cell carcinoma, and well-differentiated thyroid and oral cavity carcinoma; sarcoma; and melanoma.
* The subject is scheduled to undergo resection or biopsy of the ≥2.5 cm target tumour as a result of routine clinical treatment.
* The subject is scheduled to undergo or has received standard of care diagnostic imaging work-up (following the study centre's routine procedures), e.g. CT with or without contrast, MRI with or without contrast, bone scintigraphy, X-ray, or FDG-PET.
* Female subjects need to be either surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), post menopausal (cessation of menses for more than 1 year), or if of childbearing potential the results of a serum pregnancy test performed within 24 hours must be negative and with the result known before administration of AH-111585 (18F) Injection. Female subjects of reproductive potential should also employ an effective method of birth control. Barrier contraceptives must be used throughout the study in both sexes.
* The subject is able and willing to comply with study procedures, and signed and dated informed consent is obtained.
* The subject has a blood urea nitrogen value and serum creatinine value of ≤1.5 of the upper normal limit.
* The subject has a platelet count of >75,000 x 10^6/L.
* The subject has a haemoglobin value of >9 g/dL.
* The subject has a prothrombin time and an activated partial thromboplastin time and within normal limits.
* The subject has a clinically acceptable (as judged by the investigator) physical examination at screening and is capable of self-care, i.e. Eastern Cooperative Oncology Group performance status is 0 to 2, such that the subject has a high chance to complete the study.
* The subject has not received any anti-angiogenic agents (e.g. bevacizumab, sorafenib, sunitinib) within 10 days prior to PET imaging.
* The subject has had no open wounds within 10 days prior to study entry.
* The chosen target tumour is not within the liver.

Inclusion Criteria Specific for Subjects with High-grade Glioma:

* The subject is suspected of having supratentorial malignant primary glioma (by biopsy or presenting MRI characteristics as determined by the subject's clinician) requiring further surgical resection as part of the recommended treatment plan for their newly diagnosed disease. These gliomas include glioblastoma multiforme, anaplastic astrocytoma, and anaplastic oligodendroglioma.
* The subject has undergone recent biopsy of newly diagnosed high-grade glioma, has recovered from the effects of surgical biopsy, and baseline on-study MRI/CT is performed within 14 days of entry into the study.

Exclusion Criteria:

* The subject is lactating.
* The subject is being treated with heparin or coumadin.
* The subject has received another investigational medicinal product (IMP) within 14 days before, or will receive an IMP within 1 week after administration of AH-111585 (18F) Injection.
* The subject was previously included in this study.
* The subject experienced substantial changes in their medical status before all essential study procedures (including all imaging procedures and surgical excision or biopsy) are performed.
* The subject has any contraindication to any of the study procedures, products used or its constituents (e.g. X-ray contrast media).
* The subject has known hyper- or hypo-coagulation syndromes. Such coagulopathies include but are not limited to Von Willebrand disease, Protein C deficiency, Protein S deficiency, Hemophilia A/B/C, Factor-V Leiden, and Bernard-Soulier syndrome.
* The subject is unable to lie down for 125 minutes.
* The subject suffers from claustrophobia.
* The subject has known diagnosis of human immunodeficiency virus (HIV) infection.
* The subject has known diagnosis of hepatitis B or C infection.
* The subject has known diagnosis of mental incapacitation and it affects their ability to consent.
* The subject has been diagnosed with a primary or metastatic tumour lesion <2.5 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-11; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Winick, Ph.D., Study Director — GE Healthcare
Locations (1):
- GE Healthcare Office, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 33 subjects enrolled in this study. 16 subjects completed the study and 17 subjects did not.
Pre-assignment Details: 33 subjects enrolled,16 subjects completed and 17 did not complete. The reasons why 17 subjects that did not complete the study: 2 subjects failed screening, 6 subjects were lost to followup, 1 subject the procedure had technical problems, 2 subjects discontinued due to Physician decision, and 6 subjects had other reasons for not completing.
Groups:
- Fluciclatide Injection: The patient would receive an injection of Fluciclatide (GE-135) (F18) at 10mCi (370 megabecquerels (MBq)).
Period: Overall Study
Arm/Group | Fluciclatide Injection
Started | 33
Completed | 16
Not Completed | 17
Not completed — Screen Failure | 2
Not completed — Lost to Follow-up | 6
Not completed — Technical Problems | 1
Not completed — Physician Decision | 2
Not completed — Other reasons | 6

BASELINE CHARACTERISTICS:
Population: 33 subjects enrolled/ started the study. 25 subjects were used in this study analysis.
Groups:
- Safety With Fluciclatide Injection: The patient would receive an injection of Fluciclatide (GE-135) (F18) at 10mCi (370 megabecquerels (MBq)).
Arm/Group | Safety With Fluciclatide Injection
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (10.09)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 24
  United Kingdom | 1

OUTCOME MEASURES:

1. Primary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ3 (Beta-3 Integrin) Integrin Expression in Tumors. (Correlation Between Ki_inp-Patlak and αvβ3 Optical Density)
Description: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention by tumor tissue following intravenous administration of AH111585 (18F) Injection for the Full Analysis Set (FAS) subjects. Correlation strength was defined descriptively. 0.22 and 0.24 equals a weak positive correlation and 0.16 and 0.18 equals a negligible correlation.
  Three (3) of the 22 subjects did not have any αvβ3 integrin results. Ki-inp-Patlak is a graphical analysis technique based on the compartment model that uses linear regression to identify and analyze pharmacokinetics of tracers involving irreversible uptake.
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: This Outcome Measure was assessed among the Full Analysis Set (FAS), 3 of the 22 Subjects did not have any αvβ3 integrin results.
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between Ki_inp-Patlak and αvβ3 Optical Density: Correlation between Imaging parameters. The selected imaging parameters that reflected (18F) Fluciclatide tracer uptake and retention.
Arm/Group | Correlation Between Ki_inp-Patlak and αvβ3 Optical Density
Number analyzed (Participants) | 19
Correlation coefficient | 0.22 [-0.26 to 0.61]

2. Primary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ3 Integrin Expression in Tumors. (Correlation Between VT_inp-Logan and αvβ3 Optical Density)
Description: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention by tumor tissue following intravenous administration of AH111585 (18F) Injection for the Full Analysis Set (FAS) subjects. Correlation strength was defined descriptively.
  The Logan plot is the counterpart of the Patlak plot for reversible radiotracers.
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between VT_inp-Logan and αvβ3 Optical Density: Correlation between Imaging parameters. The selected imaging parameters that reflected (18F) Fluciclatide tracer uptake and retention.
Arm/Group | Correlation Between VT_inp-Logan and αvβ3 Optical Density
Number analyzed (Participants) | 19
Correlation coefficient | 0.24 [-0.24 to 0.62]

3. Secondary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ5 Integrin Expression in Tumors. (Correlation Between Ki_inp-Patlak αvβ5 Optical Density)
Description: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention by tumor tissue following intravenous administration of AH111585 (18F) Injection for the Full Analysis Set (FAS) subjects. Correlation strength was defined descriptively. 0.60 to 0.44 equals a moderately positive correlation and 0.33 to 0.37 equals a weak positive correlation.
  Two (2) of the 22 subjects did not have any αvβ5 integrin results.
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: This Outcome Measure was assessed among the Full Analysis Set (FAS), 2 of the 22 Subjects did not have any αvβ5 integrin results.
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between Ki_inp-Patlak αvβ5 Optical Density: The patient would receive an injection of Fluciclatide (GE-135) (F18) at 10mCi (370 megabecquerels (MBq)). Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention with Quantitative Measurement of the Levels of αvβ5 Integrin Expression in Tumors for the Full Analysis Set (FAS) subjects.
Arm/Group | Correlation Between Ki_inp-Patlak αvβ5 Optical Density
Number analyzed (Participants) | 20
Correlation coefficient | 0.60 [0.20 to 0.82]

4. Secondary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ5 Integrin Expression in Tumors. (Correlation Between VT_inp-Logan and αvβ5 Optical Density)
Description: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention by tumor tissue following intravenous administration of AH111585 (18F) Injection for the Full Analysis Set (FAS) subjects. Correlation strength was defined descriptively.
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between VT_inp-Logan and αvβ5 Optical Density: The patient would receive an injection of Fluciclatide (GE-135) (F18) at 10mCi (370 megabecquerels (MBq)). Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention with Quantitative Measurement of the Levels of αvβ5 Integrin Expression in Tumors for the Renal Cell Carcinoma (RCC) subjects.
Arm/Group | Correlation Between VT_inp-Logan and αvβ5 Optical Density
Number analyzed (Participants) | 20
Correlation coefficient | 0.44 [-0.01 to 0.73]

5. Primary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ3 (Beta-3 Integrin) Integrin Expression in Tumors. (Correlation Between SUVw_55 and αvβ3 Optical Density)
Description: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention by tumor tissue following intravenous administration of AH111585 (18F) Injection for the Full Analysis Set (FAS) subjects. Correlation strength was defined descriptively.
  SUVw_55 is the standard uptake value at 55 minutes post-injection, normalized to weight.
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between SUVw_55 and αvβ3 Optical Density: Correlation between Imaging parameters. The selected imaging parameters that reflected (18F) Fluciclatide tracer uptake and retention.
Arm/Group | Correlation Between SUVw_55 and αvβ3 Optical Density
Number analyzed (Participants) | 19
Correlation coefficient | 0.16 [-0.32 to 0.57]

6. Primary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ3 (Beta-3 Integrin) Integrin Expression in Tumors. (Correlation Between SUVR_55_blood and αvβ3 Optical Density)
Description: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention by tumor tissue following intravenous administration of AH111585 (18F) Injection for the Renal Cell Carcinoma (RCC) subjects. Correlation strength was defined descriptively.
  Twelve (12) of the 22 subjects had renal cell carcinoma (RCC) the remaining subjects did not have RCC.
  SUVR_55_blood is the standard uptake value ratio (tumor-to-blood) at 55 minutes post-injection.
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between SUVR_55_blood and αvβ3 Optical Density: Correlation between Imaging parameters. The selected imaging parameters that reflected (18F) Fluciclatide tracer uptake and retention.
Arm/Group | Correlation Between SUVR_55_blood and αvβ3 Optical Density
Number analyzed (Participants) | 19
Correlation coefficient | 0.18 [-0.30 to 0.58]

7. Primary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ3 Integrin Expression in Tumors. (Correlation Between Ki_inp-Patlak and αvβ3 Optical Density)
Description: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention by tumor tissue following intravenous administration of AH111585 (18F) Injection for the Renal Cell Carcinoma (RCC) subjects. Correlation strength was defined descriptively.
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: This Outcome Measure was assessed among the Renal Cell Carcinoma (RCC) subjects, 12 of the 22 Subjects had Renal Cell Carcinoma (RCC).
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between Ki_inp-Patlak and αvβ3 Optical Density: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention with Quantitative Measurement of the Levels of αvβ3 Integrin Expression in Tumors for the Renal Cell Carcinoma (RCC) subjects.
Arm/Group | Correlation Between Ki_inp-Patlak and αvβ3 Optical Density
Number analyzed (Participants) | 12
Correlation coefficient | 0.49 [-0.14 to 0.82]

8. Primary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ3 Integrin Expression in Tumors. (Correlation Between VT_inp-Logan and αvβ3 Optical Density)
Description: as for outcome 7
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between VT_inp-Logan and αvβ3 Optical Density: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention with Quantitative Measurement of the Levels of αvβ3 Integrin Expression in Tumors for the Renal Cell Carcinoma (RCC) subjects.
Arm/Group | Correlation Between VT_inp-Logan and αvβ3 Optical Density
Number analyzed (Participants) | 12
Correlation coefficient | 0.56 [-0.05 to 0.85]

9. Primary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ3 Integrin Expression in Tumors. (Correlation Between SUVw_55 and αvβ3 Optical Density)
Description: as for outcome 7
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between SUVw_55 and αvβ3 Optical Density: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention with Quantitative Measurement of the Levels of αvβ3 Integrin Expression in Tumors for the Renal Cell Carcinoma (RCC) subjects.
Arm/Group | Correlation Between SUVw_55 and αvβ3 Optical Density
Number analyzed (Participants) | 12
Correlation coefficient | 0.49 [-0.13 to 0.83]

10. Primary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ3 Integrin Expression in Tumors. (Correlation Between SUVR_55_blood and αvβ3 Optical Density)
Description: as for outcome 7
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between SUVR_55_blood and αvβ3 Optical Density: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention with Quantitative Measurement of the Levels of αvβ3 Integrin Expression in Tumors for the Renal Cell Carcinoma (RCC) subjects.
Arm/Group | Correlation Between SUVR_55_blood and αvβ3 Optical Density
Number analyzed (Participants) | 12
Correlation coefficient | 0.44 [-0.20 to 0.80]

11. Secondary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ5 Integrin Expression in Tumors. (Correlation Between SUVw_55 and αvβ5 Optical Density)
Description: as for outcome 4
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between SUVw_55 and αvβ5 Optical Density: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention by tumor tissue following intravenous administration of AH111585 (18F) Injection for the Full Analysis Set (FAS) subjects. Correlation strength was defined descriptively.
Arm/Group | Correlation Between SUVw_55 and αvβ5 Optical Density
Number analyzed (Participants) | 20
Correlation coefficient | 0.33 [-0.14 to 0.67]

12. Secondary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ5 Integrin Expression in Tumors. (Correlation Between SUVR_55_blood and αvβ5 Optical Density)
Description: as for outcome 4
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between SUVR_55_blood and αvβ5 Optical Density: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention by tumor tissue following intravenous administration of AH111585 (18F) Injection for the Full Analysis Set (FAS) subjects. Correlation strength was defined descriptively.
Arm/Group | Correlation Between SUVR_55_blood and αvβ5 Optical Density
Number analyzed (Participants) | 20
Correlation coefficient | 0.37 [-0.10 to 0.69]

13. Secondary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ5 Integrin Expression in Tumors. (Correlation Between Ki_inp-Patlak and αvβ5 Optical Density)
Description: as for outcome 7
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between Ki_inp-Patlak and αvβ5 Optical Density: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention by tumor tissue following intravenous administration of AH111585 (18F) Injection for the Renal Cell Carcinoma (RCC) subjects. Correlation strength was defined descriptively.
Arm/Group | Correlation Between Ki_inp-Patlak and αvβ5 Optical Density
Number analyzed (Participants) | 12
Correlation coefficient | 0.90 [0.67 to 0.97]

14. Secondary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ5 Integrin Expression in Tumors. (Correlation Between VT_inp-Logan and αvβ5 Optical Density)
Description: as for outcome 7
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between VT_inp-Logan and αvβ5 Optical Density: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention by tumor tissue following intravenous administration of AH111585 (18F) Injection for the Renal Cell Carcinoma (RCC) subjects. Correlation strength was defined descriptively.
Arm/Group | Correlation Between VT_inp-Logan and αvβ5 Optical Density
Number analyzed (Participants) | 12
Correlation coefficient | 0.78 [0.34 to 0.93]

15. Secondary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ5 Integrin Expression in Tumors. (Correlation Between SUVw_55 and αvβ5 Optical Density)
Description: as for outcome 7
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between SUVw_55 and αvβ5 Optical Density: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention by tumor tissue following intravenous administration of AH111585 (18F) Injection for the Renal Cell Carcinoma (RCC) subjects. Correlation strength was defined descriptively.
Arm/Group | Correlation Between SUVw_55 and αvβ5 Optical Density
Number analyzed (Participants) | 12
Correlation coefficient | 0.57 [-0.03 to 0.85]

16. Secondary Outcome: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention With Quantitative Measurement of the Levels of αvβ5 Integrin Expression in Tumors. (Correlation Between SUVR_55_blood and αvβ5 Optical Density)
Description: as for outcome 7
Time Frame: Tissue sample acquisition within 2 weeks of Fluciclatide PET scan.
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Correlation Between SUVR_55_blood and αvβ5 Optical Density: Correlation of the Magnitude of [18F]Fluciclatide Uptake and Retention by tumor tissue following intravenous administration of AH111585 (18F) Injection for the Renal Cell Carcinoma (RCC) subjects. Correlation strength was defined descriptively.
Arm/Group | Correlation Between SUVR_55_blood and αvβ5 Optical Density
Number analyzed (Participants) | 12
Correlation coefficient | 0.74 [0.27 to 0.92]

ADVERSE EVENTS:
Time Frame: Up to 6 weeks post administration of Fluciclatide (GE-135) (18F) Injection at 10 mCi [370 megabecquerels (MBq)].
Arm/Group | Fluciclatide Injection
Serious Adverse Events (participants affected / at risk) | 5/25
Other Adverse Events (participants affected / at risk) | 13/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluciclatide Injection (N=25)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Glioblastoma Multiforme (GBM) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Idiopathic Thrombocytopenic Purpura (ITP) (Blood and lymphatic system disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal Injury (Injury, poisoning and procedural complications) | 1 (1)
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluciclatide Injection (N=25)
Gastrointestinal Disorders (Gastrointestinal disorders) | 3 (3) — AEs were described by system organ class.
General disorders and administration site conditions (General disorders) | 5 (6) — AEs were described by system organ class.
Infections and Infestations (Infections and infestations) | 3 (3) — AEs were described by system organ class.
Investigations (Investigations) | 3 (4) — AEs were described by system organ class.
Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2) — AEs were described by system organ class.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No